CLINICAL TRIAL: NCT03866746
Title: Aflibercept With Adjuvant Micro-Pulsed Yellow Laser Versus Aflibercept Monotherapy in Treatment of Diabetic Macular Edema.
Brief Title: Aflibercept With and Without Micropulse Laser in Diabetic Macular Edema
Acronym: MPL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al Hadi Hospital (Other)
Responsible Party: Principal Investigator, Abeer MohamedSadeck Khattab, associate professor of ophthalmology, Al Hadi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlHadi Hospital
Record Dates: First submitted 2019-03-01; First posted 2019-03-07 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Macular Edema
Keywords: Aflibercept; Anti-VEGFs; micropulsed diode laser; subthreshold
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): received aflibercept injections alone
  Interventions: Drug: Aflibercept Injection
- Group B (Experimental): received 3 aflibercept injections followed by micropulsed laser
  Interventions: Drug: Aflibercept Injection; Other: micropulsed yellow laser

INTERVENTIONS:
Drug: Aflibercept Injection — Group A;Under complete aseptic conditions; intravitreal aflibercept injections with dose of 2 mg/0.05 mL per injection was given for the patients. Patients were scheduled to receive 3 loading injections at monthly interval. At the 3rd month; further treatment was planned pro re nata (PRN) according to the response. Injections were discontinued when the CMT reached 250 µm or less. If there was no change in the CMT after two consecutive injections; patients shifted to other line of treatment. Reinjection was continued for the other eyes with re-evaluation of the response every month.In group B Patients received the initial 3 monthly loading doses of IVI of aflibercept followed by MPL therapy (within one week after the 3rd injection). Patients were scheduled for follow-up monthly. Injection followed by MPL was then repeated according to the response as in group A.
  Other Names: Micropulsed yellow laser
Other: micropulsed yellow laser — Micropulse yellow IQ 577nm laser (Iridex Corporation, Mountain View, CA, USA) was employed. The Area Centralis lens (laser spot size magnification 0.94) was utilized with 400 mw power, 200μm spot size and 200 ms pulse duration with 5% duty cycle after micropulse mode activation. Laser was applied on clinically visible thickened macula with different number of confluent non- spacing shots in 7x7 grids. Care was taken to begin treatment outside the foveal avascular zone and not to treat the fovea when there was no visible reaction. If there was any visible reaction; treatment was stopped and the power was reduced until there was no visible reaction.
  Arms: Group B

SUMMARY:
prospective study evaluating the impact of subthreshold micropulsed laser on the number of Aflibercept injections when used as an adjuvant therapy in eyes with diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* diagnosed with DME with central macular thickness (CMT) more than 250 µm measured by OCT
* best corrected visual acuity (BCVA) between 20/400 and 20/40.

Exclusion Criteria:

* patients with intra-ocular surgery as cataract surgery within 6 months
* prior intravitreal injection of any drug within the preceding 6 months
* panretinal photocoagulation (PRP) within the former 4 months.
* Patients with previous macular laser
* patients with vitreo-macular traction (VMT) syndrome
* severe glaucoma
* other retinal vascular diseases
* conditions that impede the OCT interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
the number of intravitreal injections | 18th month follow-up.
  the total number of intravitreal aflibercept injections were recorded
Central macular thickness | 18 month
  in um

SECONDARY OUTCOMES:
best corrected visual acuity measured in ETDRS. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Abeer M Khattab, MD, Principal Investigator — Al Hadi Hospital
Locations (1):
- AlHadi hospital, Hawalli, AlJabryia, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided